CLINICAL TRIAL: NCT02442180
Title: Efficacy and Safety of Granulocyte-colony Stimulating Factor in Patients With Severe Alcoholic Hepatitis With Null or Partial Response to Steroid: A Randomized, Double-blind, Placebo-controlled, Nationwide Multi-center Study
Brief Title: Efficacy and Safety of G-CSF in Patients With Severe Alcoholic Hepatitis With Null or Partial Response to Steroid
Acronym: GraCiAH
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: failure to recruit eligible patients
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Dong Joon Kim, professor Dong Joon Kim, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-6
Record Dates: First submitted 2015-05-02; First posted 2015-05-13 (Estimated); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; Steroids; Prednisolone; Methylprednisolone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- G-CSF + steroid in partial responder (Experimental): Patients who are randomized to prednisolone plus G-CSF treatment group in patients with partial responder to prednisolone therapy.
  Interventions: Drug: G-CSF (Filgrastim injection); Drug: steroid
- Placebo + steroid in partial responder (Placebo Comparator): Patients who are randomized to prednisolone plus placebo treatment group in patients with partial responder to prednisolone therapy.
  Interventions: Drug: steroid; Drug: placebo
- G-CSF in null responder to steroid (Experimental): Patients who are randomized to G-CSF treatment group in patients with null responder to prednisolone therapy.
  Interventions: Drug: G-CSF (Filgrastim injection)
- Placebo in null responder to steroid (Placebo Comparator): Patients who are randomized to placebo treatment group in patients with null responder to prednisolone therapy.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: G-CSF (Filgrastim injection) — G-CSF (Filgrastim injection) 5ug/kg subcutaneous injection daily for 5 days and every 3 days (total 12 doses)
  Other Names: Filgrastim (brand name), Recombinant Filgrastim
  Arms: G-CSF + steroid in partial responder; G-CSF in null responder to steroid
Drug: steroid — oral prednisolone 40mg qd or iv methylprednisolone 32 mg if oral medication is not tolerable
  Other Names: prednisolone or methylprednisolone
  Arms: G-CSF + steroid in partial responder; Placebo + steroid in partial responder
Drug: placebo — equivalent to G-CSF doses
  Other Names: normal saline
  Arms: Placebo + steroid in partial responder; Placebo in null responder to steroid

SUMMARY:
Steroid is the treatment of choice in patients with severe alcoholic hepatitis. However, null- or partial responder of steroid treatment is recommended to consider liver transplantation. The yearly demand for liver transplants far exceeds the supply of available organs and alcoholic liver disease has been a controversial indication for transplantation. Granulocyte-Colony Stimulating Factor (G-CSF) has been reported to have effect of proliferation of hepatic progenitors in alcoholic steatohepatitis. The aim of this study is to investigate the efficacy of G-CSF in patients with severe alcoholic hepatitis with null or partial response to steroid.

DETAILED DESCRIPTION:
Severe alcoholic hepatitis is defined as alcoholic hepatitis patients having discriminant function (DF) score over 32 or accompanying hepatic encephalopathy. These patients have shown poor prognosis of 28 day mortality as 30 to 50% without treatment. Steroid (prednisolone 40mg/day for 28 days) is the treatment of choice in patients with severe alcoholic hepatitis. Alcoholic hepatitis with modified DF score greater than or equal to 32 or model for end-stage liver disease (MELD) score over 21 or with hepatic encephalopathy are indications. However, null- or partial responder of steroid treatment is recommended to consider liver transplantation. The yearly demand for liver transplants far exceeds the supply of available organs and alcoholic liver disease has been a controversial indication for transplantation. Even in the responders of steroid treatment, the mortality is still 20% (from 40% without treatment to 20% with steroid treatment). There is a need for development of new treatment for this catastrophic disease. Granulocyte-Colony Stimulating Factor (G-CSF) has been reported to have effect of proliferation of hepatic progenitors in alcoholic steatohepatitis. The aim of this study is to investigate the efficacy of G-CSF in patients with severe alcoholic hepatitis with null or partial response to steroid.

ELIGIBILITY:
Inclusion Criteria: Patients with

* Clinical significant alcohol intake history (men over 50g within 3 months, women over 40g within 3 months)
* modified DF score greater than or equal to 32
* Transjugular liver biopsy shows typical feature of alcoholic hepatitis or meet the clinical diagnosis (total serum bilirubin level over 5 mg/dL, aspartate aminotransferase/alanine aminotransferase ratio >2, aspartate aminotransferase < 300 IU/L)
* Included patients should meet the all above criteria and Lille score > 0.16 at the day 7 of prednisolone 40mg (or 32 mg of methylprednisolone) daily treatment.

Exclusion Criteria: Patients with

* hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (anti-HCV), or anti-human immunodeficiency virus (HIV) (+)
* Malignancy including hepatocellular carcinoma
* Portal vein thrombosis, hemochromatosis, autoimmune hepatitis, Wilson's disease, alpha-1-antitrypsin deficiency
* Pregnancy, breast feeding, or who refuses contraception, or who cannot do contraception
* History of adverse event including allergic response, hypersensitivity to G-CSF
* Hypovolemic shock due to gastrointestinal hemorrhage or who need packed red blood cell (RBC) transfusion more than 3 units or increased modified discriminant factor (DF) score greater or equal to 32 from below 32 due to gastrointestinal hemorrhage
* Sepsis or uncontrolled acute infection
* Hepatic encephalopathy grade 3-4
* History of steroid or pentoxifylline treatment within 3 months
* Myeloblast on peripheral blood smear test
* Critical comorbidities (type I hepatorenal syndrome, serum creatinine >2.5mg/dL, heart failure, pulmonary disease, psychiatric disease, acute pancreatitis etc.)
* Who refuses to participate in clinical trial

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
2-month survival rate of null responder to steroid treatment and 6-month survival rate of partial responder to steroid treatment | After 2 months of G-CSF or placebo treatment in patients with null responder to steroid treatment and after 6 months of G-CSF+steroid or only steroid treatment in patients with partial responder to steroid treatment
  Survival status can be determined by the occurrence of mortality regardless of any cause of death.

SECONDARY OUTCOMES:
Hepatic function improvement as assessed by the Child-Pugh score | day 0,1,3,7,9,11,14,17,20,23,26,29,32,35,60,90,120,150,180
  Hepatic function is defined as the Child-Pugh score.
Hepatic function improvement as assessed by the MELD score | day 0,1,3,7,9,11,14,17,20,23,26,29,32,35,60,90,120,150,180
  Hepatic function is defined as the MELD score.
Hepatic function improvement as assessed by the Chronic Liver Failure (CLIF)-Sequential Organ Failure Assessment (SOFA) score | day 0,1,3,7,9,11,14,17,20,23,26,29,32,35,60,90,120,150,180
  Hepatic function is defined as the CLIF-SOFA score.
Hepatic function improvement as assessed by the Fraction of Cluster of differentiation (CD34)+ cell in peripheral blood | day0,7,35
  Hepatic function is defined as the CD34+ cell count percentage in circulating blood.
Hepatic function improvement as assessed by the Alcoholic Hepatitis Histology score | day0,35
  Hepatic function is defined as histological scoring system of alcoholic hepatitis (AHHS).

CONTACTS AND LOCATIONS:
Overall Officials: Dong Joon Kim, M.D., Ph.D., Principal Investigator — Hallym Universitiy College of Medicine, Chuncheon Sacred Heart hospital, Chuncheon, South Korea
Locations (1):
- Chuncheon Sacred Heart hospital, Chuncheon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho Y, Park YS, Kim HY, Kim W, Lee HJ, Kim DJ. Efficacy of granulocyte colony stimulating factor in patients with severe alcoholic hepatitis with partial or null response to steroid (GRACIAH trial): study protocol for a randomized controlled trial. Trials. 2018 Dec 22;19(1):696. doi: 10.1186/s13063-018-3092-7. PMID 30577864